CLINICAL TRIAL: NCT06229613
Title: Exhaled Breath Aerosol for the Etiological Diagnosis of Respiratory Tract Infections: a Pilot Study
Acronym: AEROPLEX
Status: Completed | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Daniela Maria Cirillo, Head Emerging Bacterial Pathogens, IRCCS San Raffaele Scientific Institute, IRCCS Ospedale San Raffaele
Other Study IDs: AEROPLEX
Record Dates: First submitted 2023-12-22; First posted 2024-01-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Diseases
Keywords: respiratory infection; exhaled breath aerosols (XBAs); XBA collection devices
MeSH Terms: conditions — Respiratory Tract Diseases; Respiratory Tract Infections | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: medical device for exhaled breath aerosols (XBAs) collection — To evaluate the feasibility of XBAs collection and analysis (index test) using the molecular tests currently in use at San Raffaele Hospital for the detection of respiratory pathogens in clinical samples, compared to upper respiratory secretion and sputum samples, that will be collected using standard procedures and analysed using the same kits (comparator tests).

SUMMARY:
Pilot study for the evaluation of the feasibility of pathogen detection in exhaled breath aerosols (XBAs) samples using the AveloCollect device.

The aim of the study is to evaluate the feasibility of XBA collection and molecular detection of respiratory pathogens using the AveloCollect BlowTube device (index test) in subjects with a clinical presentation consistent with a respiratory infectious disease, compared to the same molecular assays performed on nasopharyngeal secretions (using commercially available swabs) and sputum (comparator tests).

DETAILED DESCRIPTION:
Respiratory infections have a significant impact in terms of morbidity and mortality, both in the EU and globally and were responsible for the majority of pandemics in the last centuries. Human breath is an attractive sample type, given the ease of sample collection via non-invasive methods, its direct link to the route of transmission, and its potential role as an indicator of infectiousness. In particular, recent studies have focused on the exhaled breath aerosols (XBAs). Aerosol transmission was demonstrated for many respiratory infections, including pandemic influenza, respiratory syncytial virus (RSV), tuberculosis (TB) and COVID-19. Pathogen detection in XBA samples has shown a good sensitivity, but currently available research tools are highly technical and resource demanding. New and simplified XBA collection devices (Face masks, AveloCollect Blow tube device) are currently under evaluation, and further clinical studies are needed in order to assess their feasibility for pathogen detection in clinical practice, especially for etiological diagnosis in patients with unspecific respiratory symptoms.

The objective of this study is to evaluate the feasibility of XBAs collection and analysis (index test) using the molecular tests currently in use at San Raffaele Hospital for the detection of respiratory pathogens in clinical samples, compared to upper respiratory secretion and sputum samples, that will be collected using standard procedures and analysed using the same kits (comparator tests).

ELIGIBILITY:
Inclusion Criteria:

* Adult age (≥18 years)
* Subjects with one or more symptoms of respiratory tract infection (fever, cough, sore throat, dyspnea, conjunctivitis and/or rhinitis).
* Samples collected within 3 days from symptom onset.
* No antibiotic drug taken during the previous 3 days

Exclusion Criteria:

* Pregnancy
* Samples collected after 3 days from symptom onset.
* Antibiotic drug taken during the previous 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare workers with fever, cough, sore throat, dyspnea, rhinitis and/or conjunctivitis will be enrolled
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of XBAs collection and analysis (index test) using the molecular tests currently in use | 8 months
  Descriptive analyses will be carried out. The samples will undergo molecular analysis in order to detect respiratory pathogens, using the tests currently in use at San Raffaele Hospital for detection of respiratory pathogens in clinical samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Emerging Bacterial Pathogens Unit, Milan, Italy, Italy